CLINICAL TRIAL: NCT04874285
Title: Supplementation With Hyaluronic Acid, Alpha-lipoic Acid, Magnesium, and Vitamin D and B6 in Patients at Risk of Abortion Treated With Progesterone: a Pilot Study.
Brief Title: Use of Dietary Supplements in Patients at Risk of Abortion Treated With Progesterone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMW-HA_ABORTION
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy, High Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Women with risk factors for abortion, treated with progesterone
- study group (Experimental): Women with risk factors for abortion, treated with progesterone and a dietary supplement containing hyaluronic acid, alpha-lipoic acid, vitamin D and vitamin B6
  Interventions: Dietary Supplement: HA

INTERVENTIONS:
Dietary Supplement: HA — hyaluronic acid, alpha-lipoic acid, vitamin D and vitamin B6
  Arms: study group

SUMMARY:
The trial aims to investigate the effect of supplementation with hyaluronic acid, alpha-lipoic acid, magnesium, vitamin D and vitamin B6 in progesterone-treated pregnant women with risk factors for abortion.

ELIGIBILITY:
Inclusion Criteria:

* Women with risk factor for abortion (sub-chorionic hematoma during gestation or ART procedures)

Exclusion Criteria:

* Other pregnancy-related conditions
* Diabetes or hypertension
* Concomitant pharmacological therapies (anticoagulant or antihypertensive)
* Use of tocolytic drugs two months prior to enrollment
* Association with hypoglycemic drugs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
reduction of the abortion rate | 1 day (single time-point before week 20 of gestation)
  rate of abortion

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Alma Res, Rome, Italy

IPD SHARING:
Plan to Share IPD: No